CLINICAL TRIAL: NCT03633630
Title: Effect of Amla Administration on Metabolic Syndrome, Insulin Sensitivity and Insulin Secretion.
Brief Title: Amla on Metabolic Syndrome, Insulin Sensitivity and Insulin Secretion
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Esperanza Martínez-Abundis, Researcher Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Amla MS
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Metabolic Syndrome
Keywords: Amla; Emblica officinalis; Metabolic Syndrome; Insulin Secretion; Insulin Sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amla (Emblica Officinalis) (Experimental): 1000 mg dose per day. Two capsules of 500 mg, one in the morning before breakfast and the other before dinner during 90 days.
  Interventions: Drug: Amla
- Placebo (Placebo Comparator): 1000 mg dose per day. Two capsules of 500 mg, one in the morning before breakfast and the other before dinner during 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amla — Capsules of 500 mg two times per day before breakfast and dinner a total dose of 1000 mg per day. During 90 days
  Other Names: Emblica Officinalis
  Arms: Amla (Emblica Officinalis)
Drug: Placebo — Capsules of 500 mg two times per day before breakfast and dinner a total dose of 1000 mg per day. During 90 days
  Other Names: Calcined Magnesia
  Arms: Placebo

SUMMARY:
Amla has demonstrated promising effects in the treatment of obesity, dyslipidemia, hypertension, insulin secretion, among others. The above mentioned findings show that Amla has an excellent potential for the prevention and treatment of metabolic syndrome.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial will be conducted in 28 patients, 30-59 years old, with diagnosis of Metabolic Syndrome according with modified International Diabetes Federation criteria. Patients will be randomly assigned to receive Amla (500mg) or homologated placebo orally twice daily, for 90 days. Before and after the intervention, the components of Metabolic Syndrome will be evaluated, waist circumference, blood pressure, levels of fasting glucose, triglycerides, cholesterol high density lipoprotein (C-HDL), total insulin secretion (Insulinogenic index), first phase of insulin secretion (Stumvoll index) and insulin sensitivity (Matsuda index).

ELIGIBILITY:
Inclusion criteria:

* Diagnosed Metabolic Syndrome according to the IDF criteria:
* - - Waist circumference: ≥80 cm (women) ≥90 cm (men), plus two or more of the following:
* - - Fasting glucose ≥ 100 mg/dL to <126 mg/dL.
* - - Triglycerides ≥150 mg/dL to <499 mg/dL
* - - HDL-C: Men ≤40 mg/dL, women ≤50 mg/dL
* - - Systolic blood pressure ≥130 to <140 mmHg
* - - Diastolic blood pressure ≥85 to <89 mmHg
* Body Mass Index between 25 and 34.9 kg/m²
* No pharmacological treatment for Metabolic Syndrome

Exclusion Criteria:

* Pregnancy or breast-feeding
* Known allergy to Amla or placebo
* History of hepatic, kidney or thyroid disease
* Drugs or supplements consumption with proven properties that modify the behavior of the Metabolic Syndrome

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Waist Circumference (WC) | 90 days
  The WC will be evaluated after an overnight fast with a flexible tape in the midpoint between the lowest rib and the iliac crest. The value will be expressed in centimeters.
Triglycerides (TGs) | 90 days
  The blood sample for determining of TGs, will be taken after an overnight fast and with a spectrophotometry method. The value will be expressed on mmol/L.
High-density Lipoprotein Cholesterol (HDL-C) | 90 days
  The blood sample for determining of HDL-C, will be taken after an overnight fast with a colorimetric method. The value will be expressed on mmol/L.
Fasting Plasma Glucose (FPG) | 90 days
  The blood sample for determining of FPG, will be taken after an overnight fast and with a spectrophotometry method. The value will be expressed on mmol/L.
Systolic Blood Pressure (SBP) | 90 days
  The SBP will be evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures will be considered as the value of SBP. The value will be expressed on mmHg.
Diastolic Blood Pressure (DBP) | 90 days
  The DBP will be evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures will be considered as the value of DBP. The value will be expressed on mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Martínez-Abundis, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics
Locations (1):
- Institute of Experimental and Clinical Therapeutics, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Athyros VG, Mikhailidis DP. High incidence of metabolic syndrome further increases cardiovascular risk in patients with type 2 diabetes. Implications for everyday practice. J Diabetes Complications. 2016 Jan-Feb;30(1):9-11. doi: 10.1016/j.jdiacomp.2015.07.012. Epub 2015 Jul 17. No abstract available. PMID 26275865
- [Background] Samson SL, Garber AJ. Metabolic syndrome. Endocrinol Metab Clin North Am. 2014 Mar;43(1):1-23. doi: 10.1016/j.ecl.2013.09.009. PMID 24582089
- [Background] Martinez-Abundis E, Mendez-Del Villar M, Perez-Rubio KG, Zuniga LY, Cortez-Navarrete M, Ramirez-Rodriguez A, Gonzalez-Ortiz M. Novel nutraceutic therapies for the treatment of metabolic syndrome. World J Diabetes. 2016 Apr 10;7(7):142-52. doi: 10.4239/wjd.v7.i7.142. PMID 27076875
- [Background] Variya BC, Bakrania AK, Patel SS. Emblica officinalis (Amla): A review for its phytochemistry, ethnomedicinal uses and medicinal potentials with respect to molecular mechanisms. Pharmacol Res. 2016 Sep;111:180-200. doi: 10.1016/j.phrs.2016.06.013. Epub 2016 Jun 15. PMID 27320046
- [Background] Akhtar MS, Ramzan A, Ali A, Ahmad M. Effect of Amla fruit (Emblica officinalis Gaertn.) on blood glucose and lipid profile of normal subjects and type 2 diabetic patients. Int J Food Sci Nutr. 2011 Sep;62(6):609-16. doi: 10.3109/09637486.2011.560565. Epub 2011 Apr 18. PMID 21495900
- [Background] Cerezo C, Segura J, Praga M, Ruilope LM. Guidelines updates in the treatment of obesity or metabolic syndrome and hypertension. Curr Hypertens Rep. 2013 Jun;15(3):196-203. doi: 10.1007/s11906-013-0337-4. PMID 23519746
- [Background] Perez-Rubio KG, Gonzalez-Ortiz M, Martinez-Abundis E, Robles-Cervantes JA, Espinel-Bermudez MC. Effect of berberine administration on metabolic syndrome, insulin sensitivity, and insulin secretion. Metab Syndr Relat Disord. 2013 Oct;11(5):366-9. doi: 10.1089/met.2012.0183. Epub 2013 Jun 28. PMID 23808999
- [Background] O'Neill S, O'Driscoll L. Metabolic syndrome: a closer look at the growing epidemic and its associated pathologies. Obes Rev. 2015 Jan;16(1):1-12. doi: 10.1111/obr.12229. Epub 2014 Nov 18. PMID 25407540
- [Background] Mendez-Del Villar M, Gonzalez-Ortiz M, Martinez-Abundis E, Perez-Rubio KG, Cortez-Navarrete M. Effect of Irvingia gabonensis on Metabolic Syndrome, Insulin Sensitivity, and Insulin Secretion. J Med Food. 2018 Jun;21(6):568-574. doi: 10.1089/jmf.2017.0092. Epub 2018 Jan 16. PMID 29336718
- [Background] Ruilope LM, Nunes Filho ACB, Nadruz W Jr, Rodriguez Rosales FF, Verdejo-Paris J. Obesity and hypertension in Latin America: Current perspectives. Hipertens Riesgo Vasc. 2018 Apr-Jun;35(2):70-76. doi: 10.1016/j.hipert.2017.12.004. Epub 2018 Feb 1. PMID 29361428
- [Background] Grundy SM. Pre-diabetes, metabolic syndrome, and cardiovascular risk. J Am Coll Cardiol. 2012 Feb 14;59(7):635-43. doi: 10.1016/j.jacc.2011.08.080. PMID 22322078
- [Background] Harano Y, Suzuki M, Koyama Y, Kanda M, Yasuda S, Suzuki K, Takamizawa I. Multifactorial insulin resistance and clinical impact in hypertension and cardiovascular diseases. J Diabetes Complications. 2002 Jan-Feb;16(1):19-23. doi: 10.1016/s1056-8727(01)00192-1. PMID 11872361
- [Background] Lim S, Eckel RH. Pharmacological treatment and therapeutic perspectives of metabolic syndrome. Rev Endocr Metab Disord. 2014 Dec;15(4):329-41. doi: 10.1007/s11154-014-9298-4. PMID 25342235
- [Background] Park SE, Park CY, Sweeney G. Biomarkers of insulin sensitivity and insulin resistance: Past, present and future. Crit Rev Clin Lab Sci. 2015;52(4):180-90. doi: 10.3109/10408363.2015.1023429. Epub 2015 Jun 4. PMID 26042993
- [Background] Gutch M, Kumar S, Razi SM, Gupta KK, Gupta A. Assessment of insulin sensitivity/resistance. Indian J Endocrinol Metab. 2015 Jan-Feb;19(1):160-4. doi: 10.4103/2230-8210.146874. PMID 25593845
- [Background] Adams-Huet B, Devaraj S, Siegel D, Jialal I. Increased adipose tissue insulin resistance in metabolic syndrome: relationship to circulating adipokines. Metab Syndr Relat Disord. 2014 Dec;12(10):503-7. doi: 10.1089/met.2014.0092. Epub 2014 Aug 27. PMID 25162912
- [Background] Krishnaveni M, Mirunalini S. Therapeutic potential of Phyllanthus emblica (amla): the ayurvedic wonder. J Basic Clin Physiol Pharmacol. 2010;21(1):93-105. doi: 10.1515/jbcpp.2010.21.1.93. PMID 20506691
- [Background] D'souza JJ, D'souza PP, Fazal F, Kumar A, Bhat HP, Baliga MS. Anti-diabetic effects of the Indian indigenous fruit Emblica officinalis Gaertn: active constituents and modes of action. Food Funct. 2014 Apr;5(4):635-44. doi: 10.1039/c3fo60366k. PMID 24577384
- [Background] Patel SS, Goyal RK, Shah RS, Tirgar PR, Jadav PD. Experimental study on effect of hydroalcoholic extract of Emblica officinalis fruits on glucose homeostasis and metabolic parameters. Ayu. 2013 Oct;34(4):440-4. doi: 10.4103/0974-8520.127731. PMID 24696584
- [Background] Usharani P, Fatima N, Muralidhar N. Effects of Phyllanthus emblica extract on endothelial dysfunction and biomarkers of oxidative stress in patients with type 2 diabetes mellitus: a randomized, double-blind, controlled study. Diabetes Metab Syndr Obes. 2013 Jul 26;6:275-84. doi: 10.2147/DMSO.S46341. Print 2013. PMID 23935377
- [Background] Yang B, Liu P. Composition and biological activities of hydrolyzable tannins of fruits of Phyllanthus emblica. J Agric Food Chem. 2014 Jan 22;62(3):529-41. doi: 10.1021/jf404703k. Epub 2014 Jan 9. PMID 24369850
- [Background] Zhang LZ, Zhao WH, Guo YJ, Tu GZ, Lin S, Xin LG. [Studies on chemical constituents in fruits of Tibetan medicine Phyllanthus emblica]. Zhongguo Zhong Yao Za Zhi. 2003 Oct;28(10):940-3. Chinese. PMID 15620182
- [Background] Vasudeva N, Yadav N, Sharma SK. Natural products: a safest approach for obesity. Chin J Integr Med. 2012 Jun;18(6):473-80. doi: 10.1007/s11655-012-1120-0. Epub 2012 Jul 22. PMID 22821661
- [Background] Kim HY, Okubo T, Juneja LR, Yokozawa T. The protective role of amla (Emblica officinalis Gaertn.) against fructose-induced metabolic syndrome in a rat model. Br J Nutr. 2010 Feb;103(4):502-12. doi: 10.1017/S0007114509991978. Epub 2009 Nov 2. PMID 19878614
- [Background] Faizal P, Suresh S, Satheesh Kumar R, Augusti KT. A study on the hypoglycemic and hypolipidemic effects of an ayurvedic drug Rajanyamalakadi in diabetic patients. Indian J Clin Biochem. 2009 Jan;24(1):82-7. doi: 10.1007/s12291-009-0014-1. Epub 2009 May 8. PMID 23105812
- [Background] Nain P, Saini V, Sharma S, Nain J. Antidiabetic and antioxidant potential of Emblica officinalis Gaertn. leaves extract in streptozotocin-induced type-2 diabetes mellitus (T2DM) rats. J Ethnopharmacol. 2012 Jun 26;142(1):65-71. doi: 10.1016/j.jep.2012.04.014. PMID 22855943
- [Background] Nazish I, Ansari SH. Emblica officinalis - Anti-obesity activity. J Complement Integr Med. 2017 Dec 5;15(2):/j/jcim.2018.15.issue-2/jcim-2016-0051/jcim-2016-0051.xml. doi: 10.1515/jcim-2016-0051. PMID 29206643
- [Background] Chen TS, Liou SY, Chang YL. Supplementation of Emblica officinalis (Amla) extract reduces oxidative stress in uremic patients. Am J Chin Med. 2009;37(1):19-25. doi: 10.1142/S0192415X09006680. PMID 19222108
- [Background] Yokozawa T, Kim HY, Kim HJ, Okubo T, Chu DC, Juneja LR. Amla (Emblica officinalis Gaertn.) prevents dyslipidaemia and oxidative stress in the ageing process. Br J Nutr. 2007 Jun;97(6):1187-95. doi: 10.1017/S0007114507691971. PMID 17506915
- [Background] Blaschke TF, Osterberg L, Vrijens B, Urquhart J. Adherence to medications: insights arising from studies on the unreliable link between prescribed and actual drug dosing histories. Annu Rev Pharmacol Toxicol. 2012;52:275-301. doi: 10.1146/annurev-pharmtox-011711-113247. Epub 2011 Sep 19. PMID 21942628